CLINICAL TRIAL: NCT03129308
Title: A Controlled Cross Sectional Study: Prevalence of Cutaneous Autoimmune Phenomena in HIV Infected Patients
Brief Title: Prevalence of Cutaneous Autoimmune Phenomena in HIV Infected Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christopher Schuster, M.D., Assoc. Prof., Medical University of Vienna
Other Study IDs: 1103/2017
Record Dates: First submitted 2017-04-07; First posted 2017-04-26 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections; Autoimmune Diseases Affecting Skin
Keywords: HIV; Cutaneous Autoantibodies; Indirect Immunofluorescence
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 4.5ml of blood will be collected per patient and serum will be stored until final processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV infected patients: 4.5 ml of blood will be collected during a routine medical check-up.
  Interventions: Diagnostic Test: Blood Sampling
- HIV negative control patients: 4.5 ml of blood will be collected during a routine medical check-up.
  Interventions: Diagnostic Test: Blood Sampling

INTERVENTIONS:
Diagnostic Test: Blood Sampling — 4.5ml of blood will be collected and analyzed for the presence of cutaneous autoantibodies (indirect immunofluorescence, desmoglein1/3, BPAG1/2, collagenVII, and envoplakin ELISA)
  Other Names: Blood Sampling in both groups

SUMMARY:
The spectrum of reported autoimmune phenomena in HIV infected patients is unexpectedly broad and - owing to the current efficacious treatment regimes - increasing. The likelihood of the occurrence of autoimmune phenomena correlates with a high CD4 count, consequently they are found most frequently soon after infection or after immune reconstitution. It is likely that recent developments, namely the recommendation to treat all patients regardless of their CD4 count, may lead to a further increase in autoimmune phenomena in HIV infected patients. In contrast to the abundance of data of rheumatological and hematological autoimmune disease in HIV infected patients, no systematic study exists which has analyzed the prevalence of autoimmune blistering disease and/or associated autoantibodies in these patients.

The investigators therefore intend to determine the prevalence of selected autoantibodies in our HIV cohort in relation to uninfected controls. According to recent guidelines, all HIV infected patients should receive anti-retroviral treatment at the earliest time point possible, making the restoration of the immune system more likely and leading to a further alignment of the life expectancy relative to age matched, uninfected controls. As a consequence, the incidence of AIBD, especially of bullous pemphigoid, for which age is the single most important risk factor, may rise.

In total, knowledge about the prevalence of AIBD specific auto antibodies might be supportive in the diagnosis of these conditions in the future.

DETAILED DESCRIPTION:
So far no systematic studies exist about the prevalence and incidence of autoimmune blistering disease (AIBD) in HIV infected patients. Various case reports have been published, though the overall frequency appears to be low. The aim of this project is to investigate the frequency of various autoantibodies specific for various AIBD such as bullous pemphigoid, epidermolysis bullosa acquisita and paraneoplastic pemphigus using commercially available ELISA (BPAG1/2, desmoglein 1/3, collagen type VII, envoplakin) as well as indirect immunofluorescence. The knowledge of the frequency of these auto-antibodies in HIV infected patients may elucidate their clinical significance and also help in the diagnosis of AIBD in HIV infected patients.

In this cross sectional study all HIV infected patients at the HIV outpatient clinic (4-Süd) of the Department of Dermatology of Vienna's Medical University will be asked to participate in this study. Currently, the cohort includes approx. 1400 HIV infected patients and it is assumed that at least 600 patients will take part. In addition, it is intended to recruit 300 HIV negative patients who wish to get tested for HIV or require counselling for post-exposure prophylaxis. After receiving the informed consent, 4.5ml of blood will be collected during a routine medical check-up and the aforementioned tests performed.

The primary outcome is the prevalence of BPAG1/2 in HIV infected patients in comparison to uninfected, age matched controls. BPAG1/2 has been chosen as the primary end point given that bullous pemphigoid has the highest frequency among all AIBD. Secondary outcome measure will encompass the prevalence of auto antibodies against desmoglein1/3, collagen type VII, envoplakin as well as results from indirect immunofluorescence studies.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* signed informed consent

Exclusion Criteria:

* unwillingness to participate in the study
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - all HIV infected patients (confirmed by ELISA, WB, and PCR) at the HIV outpatient clinic (4-Süd) of the Department of Dermatology of Vienna's Medical University
  and
  - all HIV negative patients at the HIV outpatient clinic (4-Süd) of the Department of Dermatology of Vienna's Medical University who wish to get tested for HIV or require counselling for post-exposure prophylaxis
Sampling Method: Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
prevalence of auto-antibodies against BPAG1/2 | up to 1 year
  due to the highest frequency of bullous pemphigoid among all autoimmune blistering diseases the highest differences are expected for BPAG1/2

SECONDARY OUTCOMES:
prevalence of auto-antibodies against other cutaneous antigens | up to 1 year
  prevalence of auto-antibodies against desmoglein1/3, collagenVII, envoplakin as well as results from indirect immunofluorescence studies

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Schuster, AssocProf MD, Principal Investigator — Department of Dermatology, Medical Univeristy of Vienna
Locations (1):
- Medical University of Vienna, Department of Dermatology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No